CLINICAL TRIAL: NCT00193193
Title: A Randomized, Phase II Trial of Weekly Paclitaxel, Low-Dose Estramustine, and Carboplatin Administered Either Weekly or Every Four Weeks in the Treatment of Hormone Refractory Prostate Carcinoma
Brief Title: Weekly Paclitaxel, Low-Dose Estramustine, and Carboplatin in the Treatment of Hormone Refractory Prostate Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 10
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Paclitaxel; Estramustine; Carboplatin

INTERVENTIONS:
Drug: Paclitaxel
Drug: Estramustine
Drug: Carboplatin

SUMMARY:
In this trial we will investigate how this three-drug regimen may be improved, both with respect to efficacy and toxicity, by making some modifications in the dosing and schedule in the treatment of patients with hormone refractory prostate cancer.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will receive:

Paclitaxel + Estramustine + Carboplatin

Patients will receive weekly paclitaxel and low-dose estramustine, in combination with carboplatin administered either weekly r every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate not curable with local treatment
* Disease progression while receiving hormonal therapy
* Measurable or evaluable disease
* Previous treatment with a maximum of one prior chemotherapy regimen
* ECOG performance status 0, 1, or 2.
* Adequate bone marrow, liver and kidney function
* Able to comprehend the nature of this study and give written informed consent

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* History of treatment for an invasive malignancy within five years
* Significant heart disease

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2000-08; Primary Completion 2003-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Toxicity
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC